CLINICAL TRIAL: NCT04466709
Title: The Relationship Betweensarcopenia And Myosteatosis With The Natural History Of Liver Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Manuela Merli, Professor, University of Roma La Sapienza
Other Study IDs: 5226
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Sarcopenia; Sarcopenic Obesity; Cirrhosis, Liver
Keywords: sarcopenia; myosteatosis
MeSH Terms: conditions — Sarcopenia; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: none intervention type — This is an observational study, no intervention

SUMMARY:
Malnutrition is a common figure associated with liver cirrhosis. The main component of malnutrition in liver cirrhosis is represented by sarcopenia, a condition of a progressive and generalized loss of muscle mass and strength. Many studies have reported that sarcopenia is an independent predictor of morbidity and mortality in cirrhotic patients.

Moreover, cirrhotic patients may develop simultaneous loss of skeletal muscle and gain of adipose tissue, culminating in a condition of "sarcopenic obesity".

As highlighted by a recent systematic review and meta-analysis [Van Vgut 2017] all the studies on the impact of sarcopenia/sarcopenic obesity and myosteatosis in cirrhotic patients are retrospective studies, mostly involving non-consecutive patients on the list for liver transplantation. Moreover, most of the studies were produced by non-European centers (Canadians,Americans, and Japanese) that published more papers on the same patient series. All these factors have led to a possible selection bias.

Furthermore, the methods used to evaluate sarcopenia and myosteatosis were not homogeneous (the entire muscle area, or area of the psoas or psoas diameter) as well as the cut-offs used.

For these reasons, we propose a multicentric observational prospective study aimed at analyzing the impact of sarcopenia, sarcopenic obesity and myosteatosis in cirrhotic patients not listed for liver transplantation.

Primary endpoint:

- Evaluation of the impact of sarcopenia on the mortality of cirrhotic patients not on the waiting list for liver transplantation.

Secondary end-point:

* Evaluation of the impact of sarcopenic obesity and myosteatosis on the mortality of cirrhotic patients not on the waiting list for liver transplantation.
* Evaluation of the impact of sarcopenia/sarcopenic obesity and myosteatosis on the development of complications (hepatic encephalopathy, bacterial infections, ascites, GI bleeding) in cirrhotic patients not on the waiting list for liver transplantation.
* Evaluation of the impact of sarcopenia/sarcopenic obesity and myosteatosis on the number of admissions and the days of hospitalization for such complications.
* Evaluation of the subcutaneous fat impact on mortality and morbidity of cirrhotic patients not on the waiting list for liver transplantation.
* Concordance analysis of the various methods used (different cut-off/area psoas vs. area of all muscles) for the diagnosis of sarcopenia through the analysis of CT scan.

DETAILED DESCRIPTION:
Malnutrition is a common figure associated with liver cirrhosis with an incidence ranging from 5% to 99% of patients depending on the population studied and diagnostic tools used for the diagnosis [Amodio Hepatology 2013; Merli ESPEN; Merli 2013]. Several factors are involved in the pathogenesis of malnutrition in the patient with liver cirrhosis as an inadequate dietary intake, altered nutrient uptake and alterations in the use of the substrate due to liver disease [Tandon P 2017, Plauth M 2002]. Furthermore, a variety of acute events and complications can reduce then patient's ability to take care of their food intake [Plauth M2002]. Malnutrition is associated with an increased risk of mortality, higher prevalence of portal hypertension-related complications and infections, as well as longer in hospital stay [Merli 1996, Merli 2010, Merli 2013, Tandon P Liver Transplant 2012, Montano-Loza 2012].

The main component of malnutrition in liver cirrhosis is represented by sarcopenia, a condition of a progressive and generalized loss of muscle mass and strength [Dasarathy S 2012, Montano-Loza AJ 2012, Cruz-jentoft AJ 2010]. Many studies have reported that sarcopenia is an independent predictor of morbidity and mortality in cirrhotic patients [Merli 2013, Tandon P Liver Transplant 2012, Montano-Loza 2012].

Moreover, while overweight and obesity are endemic in Western countries, these conditions have been associated with the development of chronic liver disease, worsening of liver fibrosis and progression to cirrhosis [Everhart JE 2009; Raynard B 2002]; furthermore, the body mass index(BMI) has been considered an independent risk factor for the development of decompensation among cirrhotic patients of all causes [Berzigotti A 2010].

Cirrhotic patients may develop simultaneous loss of skeletal muscle and gain of adipose tissue, culminating in a condition of "sarcopenic obesity" [Montano-Loza AJ 2016]. This observation is relevant because, despite its important role in the prognosis of cirrhosis, sarcopenia in cirrhotic patients is frequently overlooked as body composition assessments can be challenging in cirrhotic patients with fluid retention or who are overweight or frankly obese [O'Brein 2008]. In addition, muscle depletion is characterized by both a reduction in muscle size and an increased proportion of intermuscular and intramuscular fat denominated 'myosteatosis' [Montano-Loza AJ 2016]. Myosteatosis increases with age and adiposity and it is associated with metabolic abnormalities, decreased strength and mobility [Montano-Loza AJ 2016, Correa-de-Araujo R 2017].

Montano-Loza and colleagues showed that cirrhotic patients with sarcopenic obesity or myosteatosis had worse median survival compared to those patients with normal body composition [Montano- Loza A J 2016]. In previous work, Kabori et al. demonstrated an association between myosteatosis and the prevalence of diabetes mellitus in patients undergoing hepatocellular carcinoma resection [Kaibori M 2015].

Assessment of sarcopenia and myosteatosis The European Consensus Statement has identified computed tomography (CT) as the gold standard for the detection of muscle wasting in clinical trials [Cruz-Jentoft 2010] nevertheless in clinical practice, the execution of CT and MRI is difficult to be justified only for quantifying muscle mass.

However, most cirrhotic patients have imaging for surveillance of focal liver lesions, hepatocellular carcinoma, vascular disease and pre-transplant evaluation [Dasarathy 2016]. CT is more commonly used as some software enables specific tissue demarcation using precise HU thresholds [Mitsiopoulos 1998]. There is excellent reliability between different software systems, with a good reproducibility between the software package [Irving 2007]. Although heterogeneity in the literature also exists about the abdominal muscles measured (psoas or total abdominal wall) and the site of measurements (third or fourth lumbar vertebra) [Carey 2017], the measurement of the abdominal muscle area at L3-L4 is considered the gold standard due to the relative independence from the activity level and water retention [Montano-Loza 2012].

CT images have been also the most utilized as a research tool to investigate myosteatosis. It is basically assessed indirectly using muscle attenuation calculated, leading to a close correlation with direct measurements of muscle lipid content [Machann et al., 2003; Larson-Meyer et al., 2006].

Muscle radiation attenuation is a radiological characteristic that can be measured with Hounsfield units (HU) [Goodpaster et al., 2000; Goodpaster, 2002]. When muscle cross-sectional area and attenuation are reported, the most common practice is to use pre-established HU ranges to define intermuscular fat (usually -190 to -30 HU) and muscle tissue (usually -29 HU to 150 HU) [Aubrey et al., 2014].

As highlighted by a recent systematic review and meta-analysis [Van Vgut 2017] all the abovementioned studies on the impact of sarcopenia/sarcopenic obesity and myosteatosis in cirrhotic patients are retrospective studies, mostly involving non-consecutive patients on the list for liver transplantation. Moreover, most of the studies were produced by non-European centers (Canadians,Americans, and Japanese) that published more papers on the same patient series. All these factors have led to a possible selection bias.

Furthermore, the methods used to evaluate sarcopenia and myosteatosis were not homogeneous (the entire muscle area, or area of the psoas or psoas diameter) as well as the cut-offs used.

AIMS and ENDPOINT For these reasons, we propose a multicentric observational prospective study aimed at analyzing the impact of sarcopenia, sarcopenic obesity and myosteatosis in cirrhotic patients not listed for liver transplantation.

Primary endpoint:

- Evaluation of the impact of sarcopenia on the mortality of cirrhotic patients not on the waiting list for liver transplantation.

Secondary end-point:

* Evaluation of the impact of sarcopenic obesity and myosteatosis on the mortality of cirrhotic patients not on the waiting list for liver transplantation.
* Evaluation of the impact of sarcopenia/sarcopenic obesity and myosteatosis on the development of complications (hepatic encephalopathy, bacterial infections, ascites, GI bleeding) in cirrhotic patients not on the waiting list for livertransplantation.
* Evaluation of the impact of sarcopenia/sarcopenic obesity and myosteatosis on the number of admissions and the days of hospitalization for such complications.
* Evaluation of the subcutaneous fat impact on mortality and morbidity of cirrhotic patients not on the waiting list for liver transplantation.
* Concordance analysis of the various methods used (different cut-off/area psoas vs. area of all muscles) for the diagnosis of sarcopenia through the analysis of CT scan.

PATIENTS Collection of a large national cohort of patients with liver cirrhosis not listed for liver transplantation, undergoing CT-scan abdomen based on different indications (with or without contrast). Each center needs to enroll at least 10 patients within 6 months for an estimate of at least 20 participating Italian centers.

INCLUSION CRITERIA: all patients with liver cirrhosis (age 40 - 75 years) undergoing abdominal CT-scan including the third lumbar L3 vertebrae for the clinical indication (surveillance of focal liver lesions, vascular evaluation, pre-transplant evaluation, pre-TIPS evaluation.) will be considered for the enrollment.

ELIGIBILITY:
Inclusion Criteria:

all patients with liver cirrhosis (age 40 - 75 years) undergoing abdominal CT-scan including the third lumbar L3 vertebrae for the clinical indication (surveillance of focal liver lesions, vascular evaluation, pre-transplant evaluation, pre-TIPS evaluation.) will be considered for the enrollment.

Exclusion Criteria:

1. Active list for liver transplantation (LT) (patients at evaluation for LT will beenrolled);
2. hepatocellular carcinoma HCC;
3. previous LT or listing for multivisceral or living-related LT;
4. concomitant neuromuscular disease;
5. Patients with acute or subacute liver failure without underlying cirrhosis;
6. Evidence of current malignancy except for non-melanocytic skin cancer;
7. Presence or history of severe extra-hepatic diseases (e.g., chronic renal failure requiring hemodialysis, severe heart disease (NYHA III-IV); severe chronic pulmonary disease (GOLD > III), severe neurological and psychiatric disorders);
8. HIV-positive patients;
9. Patients who decline to participate or who cannot provide prior written informed consent and when there is documented evidence that the patient has no legal surrogate decision maker and it appears unlikely that the patient will regain consciousness or sufficient ability to provide delayed informed consent;

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample size has been planned using results from an analogous retrospective study, where the HR for sarcopenia was estimated as 2.2, the 1-y event rate was 30%, and 40% of the sample had sarcopenia. We therefore conservatively assume a sHR equal to 2, 20% 1-y cause-specific event rate, 40% baseline sarcopenia. According to these data, a total of 68 cause-specific events are needed to guarantee the power of at least 80% with a type I error rate of 5%. Since we assume a 20% event rate, with a follow-up of 1y as planned 340 patients (68/0.2) will be enrolled. Considering a possible 10% drop-out, a total of 374 patients will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 374 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2020-07-05 (Actual); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
sarcopenia and mortality | 1 year
  Evaluation of the impact of sarcopenia on the mortality of cirrhotic patients not on the waiting list for liver transplantation.

SECONDARY OUTCOMES:
sarcopenic obesity/myosteatosis and mortality | 1 year
  Evaluation of the impact of sarcopenic obesity and myosteatosis on the mortality of cirrhotic patients not on the waiting list for liver transplantation.
sarcopenia, sarcopenic obesity/myosteatosis and complication of liver disease | 1 year
  Evaluation of the impact of sarcopenia/sarcopenic obesity and myosteatosis on the development of complications (hepatic encephalopathy, bacterial infections, ascites, GI bleeding) in cirrhotic patients not on the waiting list for livertransplantation.
Methods Concordance | 1 year
  Concordance analysis of the various methods used (different cut-off/area psoas vs. area of all muscles) for the diagnosis of sarcopenia through the analysis of CT scan.

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Merli, Professor, Principal Investigator — Sapeinza University of Roma
Locations (1):
- Gastroenterology Department, Sapienza University of Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No